CLINICAL TRIAL: NCT05292365
Title: Respiratory Exacerbation Plans for Action and Care Transitions for Children With Severe Cerebral Palsy (CP)
Brief Title: Respiratory Exacerbation Plans for Action and Care Transitions for Children With Severe CP
Acronym: RE-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-1532; R34HL153570-01A1 (NIH); A536771 (Other: UW Madison); Protocol Version 2/24/2023 (Other: UW Madison)
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy
Keywords: caregiver; support
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: eligible caregiver/child dyads are randomized to intervention or active control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RE-PACT Intervention (Experimental): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  Interventions: Behavioral: RE-PACT Intervention
- Active Control (AC) (No Intervention): AC subjects will receive usual comprehensive medical care and coordination.

INTERVENTIONS:
Behavioral: RE-PACT Intervention — * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  Arms: RE-PACT Intervention

SUMMARY:
This study will pilot test a just-in-time (JIT) adaptive intervention to reduce severe respiratory illness, for children with severe cerebral palsy (CP). The intervention program, called RE-PACT, delivers timely, customized action planning and health coaching when mobile text messaging with families predicts hospitalization risk is elevated. A total of n=90 caregivers of children with severe CP will be enrolled from the University of Wisconsin-Madison (UW) and the University of California, Los Angeles (UCLA) and can expect to be on study for up to 6 months.

DETAILED DESCRIPTION:
The two-site study takes place at clinical programs at US children's hospitals: the UW and UCLA Pediatric Complex Care Pro-grams were each established to deliver care to children with medical complexity. Each program is comprised of primary care providers, care coordinators, and extended visit lengths, deliver comprehensive care to children with cerebral palsy. These sites have existing collaborative relationships through their participation in the CYSHCNet national research network (http://cyshcnet.org) and other federally funded initiatives, and a track record of successful productive scientific collaboration.

The study period will be divided into three waves: after each wave, feasibility, acceptability, and fidelity data will be reviewed against pre-defined measures of success to adjust the protocol and overcome implementation barriers.

This study will be conducted through a six-month randomized pilot trial. Briefly, after recruitment and baseline assessments, eligible caregiver/child dyads are randomized to intervention (I) or active control (AC). Intervention subjects receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted. AC subjects will receive usual comprehensive medical care and coordination. Assessments of feasibility, acceptability and fidelity, as well as clinical outcomes, will be conducted at baseline and monthly intervals for 6 months. Intervention outcomes will be evaluated at baseline (i.e., randomization) and 6 months post-enrollment, and will also include the primary clinical outcome (i.e., hospitalization for respiratory diagnosis).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Primary caregiver to an eligible child (child criteria below)
* Speak English or Spanish well enough to be interviewed
* Have a phone capable of sending/receiving text messages
* Has a child

  * age 0-17 years
  * with Gross Motor Function Classification System level IV or V Cerebral Palsy
  * Cared for by respiratory specialist or receive daily respiratory treatments (oxygen, ventilation, airway clearance device, medications)

Exclusion Criteria:

* Lack of interest in text messaging or coaching interactions during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Coller, MD, MPH, Principal Investigator — UW School of Medicine and Public Health
Locations (2):
- United States (2):
  - University of California, Los Angeles, California
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
  Data prepared for distribution under a data-use agreement will be redacted to ensure privacy of study participant identity. The data-use agreement will include requirements to protect participants' privacy and data confidentiality. It will prohibit the recipient from transferring the data to other users and require that the data's security be protected by standard means and be used for research purposes only.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint analyses by contacting the study PI.
Access Criteria: The method of distribution will be by request to the study PI. After review and approval, a requestor completes the data-sharing agreement, requestor will receive a limited dataset mailed by CD or emailed through UW-Madison secured email systems that require users to create an account and sign-in with a username and password in order to receive and download any type of sensitive data.

REFERENCES:
- [Derived] Coller RJ, Singh-Verdeflor K, Eickhoff J, Chung PJ, Kloster HM, Cushing CC, Gerber DM, Katz BJ, Ia S, Wagner T, Delgado-Martinez R, Warner G, Porras-Javier L, Klitzner TS, Lerner CF. Preventing respiratory illness in cerebral palsy: Results of a pilot randomized controlled trial. PLoS One. 2025 Jun 16;20(6):e0325970. doi: 10.1371/journal.pone.0325970. eCollection 2025. PMID 40522978
- [Derived] Fleischman A, Lerner C, Kloster H, Chung P, Klitzner T, Cushing C, Gerber D, Katz B, Warner G, Singh-Verdeflor KD, Delgado-Martinez R, Porras-Javier L, Ia S, Wagner T, Ehlenbach M, Coller R. Adaptive Intervention to Prevent Respiratory Illness in Cerebral Palsy: Protocol for a Feasibility Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Jan 8;13:e49705. doi: 10.2196/49705. PMID 38190242

RESULTS

PARTICIPANT FLOW:
Groups:
- RE-PACT Intervention: Child; RE-PACT Intervention: Caregiver: Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention:
  * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
- Active Control (AC): Child; Active Control (AC): Caregiver: AC subjects will receive usual comprehensive medical care and coordination.
Period: Overall Study
Arm/Group | RE-PACT Intervention: Child | RE-PACT Intervention: Caregiver | Active Control (AC): Child | Active Control (AC): Caregiver
Started | 36 (Children were enrolled as caregiver/child dyads where caregiver n = 35 and child n = 36. One caregiver enrolled two children.) | 35 | 24 (Children were enrolled as caregiver/child dyads where caregiver n = 24 and child n = 24.) | 24
Completed | 35 | 34 | 24 | 24
Not Completed | 1 | 1 | 0 | 0
Not completed — Met Exclusion Criteria: Participant disenrolled from their complex care program | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RE-PACT Intervention: Child | RE-PACT Intervention: Caregiver | Active Control (AC): Child | Active Control (AC): Caregiver | Total
Number analyzed (Participants) | 36 | 35 | 24 | 24 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36 | 0 | 24 | 0 | 60
  Between 18 and 65 years | 0 | 35 | 0 | 24 | 59
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Per the planned analyses, totals were calculated separately for participants in the caregiver and child groups Population: Per the planned analyses, totals were calculated separately for participants in the caregiver and child groups
  years
    Child: number analyzed (Participants) | 36 | 0 | 24 | 0 | 60
    Child | 11 [5 to 14.5] |  | 9 [6 to 12] |  | 10 [5 to 14]
    Caregiver: number analyzed (Participants) | 0 | 35 | 0 | 24 | 59
    Caregiver |  | 42 [37 to 48] |  | 37 [34 to 42] | 40 [35 to 46]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data due to non-response
  Participants
    number analyzed (Participants) | 36 | 35 | 22 | 22 | 115
    Female | 10 | 32 | 11 | 22 | 75
    Male | 26 | 3 | 11 | 0 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 9 | 7 | 39
  Not Hispanic or Latino | 22 | 21 | 12 | 15 | 70
  Unknown or Not Reported | 3 | 2 | 3 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 3 | 10
  White | 26 | 25 | 12 | 15 | 78
  More than one race | 3 | 2 | 2 | 1 | 8
  Unknown or Not Reported | 3 | 4 | 7 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 36 | 35 | 24 | 24 | 119

OUTCOME MEASURES:

1. Primary Outcome: Feasibility: Number of Days to Meet Target Enrollment Size
Description: Feasibility will, in part, be measured by the number of days to meet target enrollment by wave. There are a total of 3 recruitment waves.
  This Outcome Measure was assessed by child.
Time Frame: up to 3 months
Population: *Recruitment duration was not stratified by arm.
Measure: Number; unit: Days
Groups:
- RE-PACT Intervention + Active Control (AC): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention:
  * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  AC subjects will receive usual comprehensive medical care and coordination.
  *Recruitment duration was not stratified by arm.
Arm/Group | RE-PACT Intervention + Active Control (AC)
Number analyzed (Participants) | 60
Days
  Wave 1: number analyzed (Participants) | 10
  Wave 1 | 56
  Wave 2: number analyzed (Participants) | 20
  Wave 2 | 29
  Wave 3: number analyzed (Participants) | 30
  Wave 3 | 129

2. Primary Outcome: Feasibility: Median Number of Days Between Randomization and Intervention Activities
Description: Feasibility will, in part, be measured by the number of days between randomization and (time zero) intervention activities.
  This Outcome Measure was assessed by child.
Time Frame: up to 3 months
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- RE-PACT Intervention: Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention:
  * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Days | 4 [3.5 to 7]

3. Primary Outcome: Feasibility: Mean Number of Minutes Logged for Action Planning
Description: Feasibility will, in part, be measured by the amount of time it takes to deliver the intervention.
  This Outcome Measure was assessed by child.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- RE-PACT Intervention: Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention: • Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Minutes | 22.8 (10.9)

4. Primary Outcome: Feasibility: Mean Number of Minutes Logged for Clinical Response / Coaching
Description: as for outcome 3
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Minutes | 86.8 (122.2)

5. Primary Outcome: Feasibility: Mean Number of Intervention Triggers Per Patient
Description: Feasibility will, in part, be measured by the number of intervention triggers per patient (annualized), including respiratory and non-respiratory triggers.
  This Outcome Measure was assessed by child.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Intervention Triggers
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Intervention Triggers | 0.7 (1)

6. Primary Outcome: Feasibility: Incidence of Data Infrastructure Issues
Description: Feasibility will in part be measured by the presence of necessary data infrastructure issues. This is a measure of the presence of complete data collection, between 2 sites, data use agreements and Institutional Review Board reliance. This outcome includes any events that occur over the study duration.
Time Frame: up to 22 months
Population: Number analyzed represents the number of participants by wave.
Measure: Number; unit: Data Infrastructure Issues
Groups:
- RE-PACT Intervention + Active Control (AC): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention:
  * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  AC subjects will receive usual comprehensive medical care and coordination.
  *Data Infrastructure issues were not stratified by arm.
Arm/Group | RE-PACT Intervention + Active Control (AC)
Number analyzed (Participants) | 60
Data Infrastructure Issues
  Wave 1: number analyzed (Participants) | 10
  Wave 1 | 0
  Wave 2: number analyzed (Participants) | 20
  Wave 2 | 0
  Wave 3: number analyzed (Participants) | 30
  Wave 3 | 0

7. Primary Outcome: Acceptability: Participant Enrollment Rate
Description: Acceptability will in part be measured by the participant enrollment rate, or the number of participants enrolled divided by the number of participants approached + potentially eligible.
  This Outcome Measure was assessed by child.
Time Frame: up to 6 months
Population: The number of participants analyzed must reflect the number of participants approached in addition to those consented. Enrollment rate was not stratified by arm.
Measure: Count of Participants; unit: Participants
Groups:
- RE-PACT Intervention + Active Control (AC): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention: • Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  AC subjects will receive usual comprehensive medical care and coordination.
  *Recruitment rate was not stratified by arm.
Arm/Group | RE-PACT Intervention + Active Control (AC)
Number analyzed (Participants) | 149
Participants | 60

8. Primary Outcome: Acceptability: Categorized Reasons for Consent Refusal
Description: Acceptability will in part be assessed by collecting potential participants reason for not consenting to the study. Reasons will be summarized in tabular form.
  This Outcome Measure was assessed in caregivers.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Individuals Approached for Study Recruitment: A total of 193 individuals were approached for recruitment.
Arm/Group | Individuals Approached for Study Recruitment
Number analyzed (Participants) | 133
Participants
  Ineligible: Does not have Cerebral Palsy | 9
  Ineligible: Does not meet motor function criteria | 10
  Ineligible: Does not receive respiratory care | 16
  Ineligible: Not enrolled in a complex care program | 6
  Ineligible: Moving out of the area | 1
  Ineligible: Does not meet English or Spanish language proficiency | 2
  Recruitment completed before enrollment | 4
  Not interested in the intervention | 35
  Not interested in research | 5
  Too busy | 7
  Unable to contact | 38

9. Primary Outcome: Acceptability: Participant Drop Out Rate
Description: Acceptability will in part be measured by the participant drop out rate.
  This Outcome Measure was assessed by child.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 36 | 24
Participants
  Completed Intervention | 35 | 24
  Dropped-out | 1 | 0

10. Primary Outcome: Acceptability: Measured by Mean Number of Months Participants Reported Using Action Plan
Description: Acceptability of the intervention will in part be measured by the participant feedback.
  - The number of months, on average, where participants reported use of an action plan.
  This Outcome Measure was assessed by dyad.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Months | 1.6 (1.6)

11. Primary Outcome: Acceptability: Measured by Number of Participants Reporting Definite or Probably About Recommendation of Action Plan to Others
Description: Acceptability of the intervention will in part be measured by the participant feedback.
  - Number of participants reporting definite or probably recommendation of action planning to others.
  This Outcome Measure was assessed by dyad.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 35
Participants
  Probably or Definitely recommends action planning to others | 25
  Possibly, Probably not, or Definitely does not recommend action planning to others | 10

12. Primary Outcome: Acceptability: Measured by Number of Participants Reporting Definite or Probably About Recommendation of Texting and Clinical Response to Others
Description: Acceptability of the intervention will in part be measured by the participant feedback.
  - Number of participants reporting definite or probably recommendation of texting and clinical response to others.
  This Outcome Measure was assessed in dyads.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 35
Participants
  Probably or Definitely recommends testing and/or clinical response to others | 27
  Possibly, Probably not, or Definitely does not recommend testing and/or clinical response to others | 8

13. Primary Outcome: Acceptability: Measured by Number of Participants Reporting Definite or Probably About Whether to Continue Intervention After Study is Done
Description: Acceptability of the intervention will in part be measured by the participant feedback.
  - 'How much would you want these approaches to continue as a part of regular care after the study is done?'.
  This Outcome Measure was assessed in dyads.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 35
Participants
  Probably or Definitely wants these approaches to continue as a part of regular care | 23
  Possibly, Probably not, or Definitely does not want approaches to continue as a part of regular care | 12

14. Primary Outcome: Acceptability: System Usability Scale - Composite Score
Description: Acceptability of the intervention will in part be measured by composite score. The System Usability Scale is a 10-item survey scored on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher usability. Score range = 0 - 100.
  This Outcome Measure was assessed in dyads.
  To calculate the score:
  Step 1: Convert the scale into number for each of the 10 questions Strongly Disagree: 1 point Disagree: 2 points Neutral: 3 points Agree: 4 points Strongly Agree: 5 points
  Step 2: Calculate X = Sum of the points for all odd-numbered questions - 5 Y = 25 - Sum of the points for all even-numbered questions SUS Score = (X + Y) x 2.5
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 35
score on a scale | 79.5 (11.7)

15. Primary Outcome: Fidelity: Time of Participant Enrollment in the Study
Description: Fidelity of the intervention will in part be measured by the amount of time (in months) the participant was enrolled in the study. The target participation time is 6 months.
  This Outcome Measure was assessed in children.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 36 | 24
Months | 5.9 (0.5) | 6 (0)

16. Primary Outcome: Fidelity: Number of Respiratory Action Plans Per Patient
Description: Fidelity of the intervention will in part be measured by the number of respiratory and overall action plans per patient. The goal is greater than or equal to 1.
  This Outcome Measure was assessed in children.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Respiratory Action Plans
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Respiratory Action Plans | 1 (0)

17. Primary Outcome: Fidelity: Number of Overall Action Plans Per Patient
Description: as for outcome 16
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: Overall Action Plans
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Overall Action Plans | 1 (0)

18. Primary Outcome: Fidelity: Coaching Visit Success Rate by Intervention Trigger
Description: Fidelity of the intervention will in part be measured by the coaching visit success rate, which is the number of visits (at home or virtually) completed divided by the number of visits expected), stratified by trigger. The goal is over 80 percent.
  This Outcome Measure was assessed in children.
Time Frame: up to 6 months
Population: Rows are stratified by trigger type. There are 26 triggers total, of which n = 9 are due to caregiver confidence, n = 9 are due to hospital discharge, n = 4 are due to caregiver contact, and n = 4 are due to multiple triggers.
Measure: Count of Units; unit: Intervention triggers
Units Other Than Participants: Intervention triggers
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 17
Number analyzed (Intervention triggers) | 26
Intervention triggers
  Trigger: Caregiver reported confidence < 5: number analyzed (Intervention triggers) | 9
  Trigger: Caregiver reported confidence < 5: Clinical response completed for trigger | 9
  Trigger: Caregiver reported confidence < 5: Clinical response NOT completed for trigger | 0
  Trigger: Hospital Discharge: number analyzed (Intervention triggers) | 9
  Trigger: Hospital Discharge: Clinical response completed for trigger | 9
  Trigger: Hospital Discharge: Clinical response NOT completed for trigger | 0
  Trigger: Caregiver calls or messages complex care team: number analyzed (Intervention triggers) | 4
  Trigger: Caregiver calls or messages complex care team: Clinical response completed for trigger | 4
  Trigger: Caregiver calls or messages complex care team: Clinical response NOT completed for trigger | 0
  Trigger: Multiple triggers: number analyzed (Intervention triggers) | 4
  Trigger: Multiple triggers: Clinical response completed for trigger | 4
  Trigger: Multiple triggers: Clinical response NOT completed for trigger | 0

19. Primary Outcome: Fidelity: Coaching Phone Call Success Rate by Intervention Trigger - Caregiver Reported Confidence < 5
Description: Fidelity of the intervention will in part be measured by the coaching phone call completion rate, which is the number of calls completed divided by the number of calls expected), stratified by trigger. The goal is over 80 percent.
  This Outcome Measure was assessed in children.
Time Frame: up to 6 months
Population: More follow-ups were completed than expected.
Measure: Number; unit: Follow-Ups
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 5
Follow-Ups
  Number completed | 20
  Number expected | 18

20. Primary Outcome: Fidelity: Coaching Phone Call Success Rate by Intervention Trigger - Hospital Discharge
Description: as for outcome 19
Time Frame: up to 6 months
Population: More follow-ups were completed than expected.
Measure: Number; unit: Follow-Ups
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 5
Follow-Ups
  Number completed | 30
  Number expected | 18

21. Primary Outcome: Fidelity: Coaching Phone Call Success Rate by Intervention Trigger - Caregiver Calls or Messages Complex Care Team
Description: as for outcome 19
Time Frame: up to 6 months
Population: More follow-ups were completed than expected.
Measure: Number; unit: Follow-Ups
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 4
Follow-Ups
  Number completed | 9
  Number expected | 8

22. Primary Outcome: Fidelity: Coaching Phone Call Success Rate by Intervention Trigger - Multiple Triggers
Description: as for outcome 19
Time Frame: up to 6 months
Population: More follow-ups were completed than expected.
Measure: Number; unit: Follow-Ups
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 3
Follow-Ups
  Number completed | 10
  Number expected | 8

23. Primary Outcome: Fidelity: Text Message Response Rate
Description: Fidelity of the intervention will in part be measured by the response rate to mHealth text messages, which is the number of texts responded divided by the number of texts expected.
  This Outcome Measure was assessed in dyads.
Time Frame: up to 6 months
Measure: Number; unit: Text messages
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Text messages
  Number completed | 867
  Number expected | 889

24. Primary Outcome: Fidelity: Number of Participants Inappropriately Receiving Intervention
Description: Fidelity of the intervention will in part be measured by cross-over, which is the number of participants inappropriately receiving the intervention component.
  This Outcome Measure was assessed in children.
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 36 | 24
Participants | 0 | 0

25. Primary Outcome: Fidelity: Data Collection Rate: Enrollment Surveys
Description: Fidelity of the intervention will in part be measured by the data collection rate, which is the number of data collection events complete divided by the number of total data collections events possible.
  This Outcome Measure was assessed in dyads.
Time Frame: Baseline to 2 months
Population: *Data collection was not stratified by arm.
Measure: Number; unit: Completed Enrollment Surveys
Groups:
- RE-PACT Intervention + Active Control (AC): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention:
  * Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  AC subjects will receive usual comprehensive medical care and coordination.
Arm/Group | RE-PACT Intervention + Active Control (AC)
Number analyzed (Participants) | 60
Completed Enrollment Surveys | 59

26. Primary Outcome: Fidelity: Data Collection Rate: Monthly Surveys
Description: as for outcome 25
Time Frame: up to 6 months
Measure: Number; unit: Completed Monthly Surveys
Units Other Than Participants: Monthly surveys
Groups:
- RE-PACT Intervention: Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention: • Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
    * Only intervention participants received monthly surveys.
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
Number analyzed (Monthly surveys) | 216
Completed Monthly Surveys | 210

27. Primary Outcome: Fidelity: Data Collection Rate: Exit Surveys
Description: as for outcome 25
Time Frame: up to 6 months
Population: *Data collection was not stratified by arm.
Measure: Number; unit: Completed Exit Surveys
Groups:
- RE-PACT Intervention + Active Control (AC): Intervention participants receive respiratory illness action plans and weekly mobile health (mHealth) confidence surveillance. At times of low confidence or hospitalization, just-in-time action planning and coaching activities are conducted.
  RE-PACT Intervention: • Create respiratory illness action plan
  * Weekly mHealth text messages
  * Monthly study assessments
  * Action planning and JIT coaching
  AC subjects will receive usual comprehensive medical care and coordination.
  *Data collection was not stratified by arm.
Arm/Group | RE-PACT Intervention + Active Control (AC)
Number analyzed (Participants) | 59
Completed Exit Surveys | 55

28. Secondary Outcome: Incidence of Respiratory Diagnosis Requiring Hospitalization
Description: Severe respiratory illness, defined as respiratory diagnoses requiring hospitalization. Respiratory diagnoses includes discharge diagnosis of any of the following: asthma, pneumonia (community or hospital acquired), bronchiolitis, influenza, upper or lower respiratory tract infection, tracheitis, aspiration pneumonia/pneumonitis, chronic lung disease, respiratory failure.
  - Number of children with at least 1 severe respiratory illness
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Participants
  Children with at least one severe respiratory illness | 8 | 11
  Children with no severe respiratory illness | 18 | 13

29. Secondary Outcome: Total Hospital Days During Severe Respiratory Illness by Arm
Description: Hospital days were summed by arm.
Time Frame: up to 6 months
Measure: Number; unit: Hospital Days
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Hospital Days | 8 | 32

30. Secondary Outcome: Number of Systemic Steroid Courses
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Participants
  Children with at least one systemic steroid course | 3 | 3
  Children with no systemic steroid course | 23 | 21

31. Secondary Outcome: Number of Systemic Antibiotic Courses
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Participants
  Children with at least one systemic antibiotic course throughout the study time frame | 5 | 6
  Children with no systemic antibiotic course throughout the study time frame | 21 | 18

32. Secondary Outcome: Number of Respiratory Emergency Department Visits
Time Frame: up to 6 months
Measure: Number; unit: Respiratory ED Visits
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Respiratory ED Visits | 0 | 3

33. Secondary Outcome: Child Mortality Rate
Time Frame: up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 26 | 24
Participants
  Child death | 0 | 0
  No child death | 26 | 24

34. Other Pre Specified Outcome: Family Caregiver Activation in Transition Measure (FCAT) - Mean Composite Score
Description: Capability is in part measured by the FCAT mean composite score,. FCAT is a 10-item survey to assess the caregiver's challenges on the day it is taken, scored on a 5 point likert scale from 1 (disagree strongly) to 5 (agree strongly). The mean composite score ranges from 1 - 5 with higher scores indicating higher activation. Activation of a family member refers to their desire, knowledge, confidence, and skills that can inform engagement in healthcare.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 34 | 21
score on a scale | 4.5 (0.4) | 4.5 (0.4)

35. Other Pre Specified Outcome: Caregiver General Self-Efficacy Scale (GSES) - Sum Composite Score
Description: Capability is in part measured by the GSES sum composite score. GSES is a 10-item survey scored on a 4-point Likert scale from 1 (not true at all) to 4 (exactly true). The sum composite score ranges from 10 - 40, with higher scores indicating higher efficacy.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 33 | 20
score on a scale | 34.2 (4.4) | 35.3 (4.2)

36. Other Pre Specified Outcome: Family Experiences With Care Coordination (FECC): Care Coordination Question Set
Description: Opportunity is assessed via the FECC score, using measure specifications for each item(s). The Care Coordination Question set assesses the statement "Care Coordinator Was Knowledgeable, Supportive and Advocated for Child's Needs" on a scale from 0 - 100 with
  * 0 = "Care Coordinator Was NOT Knowledgeable, Supportive and Advocated for Child's Needs"
  * 100 = "Care Coordinator Was DEFINITELY Knowledgeable, Supportive and Advocated for Child's Needs."
  This Outcome Measure was assessed in dyads.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RE-PACT Intervention | Active Control (AC)
Number analyzed (Participants) | 35 | 24
score on a scale | 87.3 (19.1) | 94.2 (8.2)

37. Other Pre Specified Outcome: Average Confidence Responses Reported by mHealth Texting
Description: Motivation is assessed by the confidence response to weekly texting and averaged over time by participant. (1-10 with higher scores indicating increased confidence).
  This Outcome Measure was assessed in dyads.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RE-PACT Intervention
Number analyzed (Participants) | 36
score on a scale | 8.59 (1.62)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during active study participation (from 4/14/2022 to 2/14/2024); any reportable events are followed to completion. Participants were assessed from enrollment to study exit, an average of six months. Caregivers were not followed for adverse events.
Description: Per protocol, information indicating an undesirable experience with study participation was reported to PI to determine if it's associated with the study. Associated events were reported to the IRB per local guidelines: https://irb.wisc.edu/wp-content/uploads/sites/2/sites/2/2022/07/AEdecisionguidewithFDAVAupdate_10_31_17.pdf. Additionally, events are documented in study files as Note-to-File. All SAEs and study-associated AEs are reported. Non-study related AEs were not collected or reported.
Arm/Group | RE-PACT Intervention | Active Control (AC)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/24
Other Adverse Events (participants affected / at risk) | 0/36 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RE-PACT Intervention (N=36) | Active Control (AC) (N=24)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT05292365/Prot_SAP_001.pdf
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT05292365/ICF_000.pdf